CLINICAL TRIAL: NCT03050502
Title: The Management of Traumatic Hemothoraces in Blunt Thoracic Injured Patients: A Randomized Clinical Trial
Brief Title: The Management of Traumatic Hemothoraces
Acronym: HemoTxRCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Principal Investigator, Dr. Chad G. Ball, Associate Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB16-1056
Record Dates: First submitted 2017-02-02; First posted 2017-02-13 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Hemothorax; Thoracic Injuries
Keywords: Hemothorax; Management
MeSH Terms: conditions — Hemothorax; Thoracic Injuries | interventions — Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chest tube drain (Active Comparator): A chest tube placed with the intent of draining all intra-pleural blood.
  Interventions: Device: Chest tube drain
- Expectant management (Sham Comparator): No chest tube, but will undergo standard observation/conservative management by the trauma service.
  Interventions: Other: Expectant management

INTERVENTIONS:
Device: Chest tube drain — This group will have an intra-pleural catheter placed with the intent of draining all intra-pleural blood (HTX). The size and nature of the catheter, manner of placement, and timing of removal will be at the discretion of the attending clinician.
  Arms: Chest tube drain
Other: Expectant management — This group will not have an intra-pleural catheter placed on the basis of the HTX, but will undergo standard observation/conservative management by the trauma service. Intra-pleural catheters may be placed after enrollment at the attending clinician's discretion.
  Arms: Expectant management

SUMMARY:
Chest injuries are common in patients with polytrauma and are responsible for approximate 25% of all trauma-related mortalities. Traumatic injuries to the thorax often result in the accumulation of blood within the chest (i.e. a hemothorax (HTX)). The management of HTX remains a clinical dilemma when the volume of blood is small to moderate and the patient is hemodynamically stable. The East American Association of Trauma guidelines suggest that all HTXs should be considered for chest tube drainage. However, a prospective observational study suggested small to moderate HTXs could be absorbed without intervention. Although HTXs are effectively managed with chest tube drainage of the blood (i.e. tube thoracostomy), this intervention is associated with numerous potential major complications, including injury and infection in up to 22% of patients. The purpose of this study is therefore to conduct a randomized controlled study to compare patients with traumatic HTX managed by chest tube drain or expectant management (close monitoring), to determine when a chest tube is needed and when it is not to treat hemothoraces. The results from this study will inform the care of future trauma patients who present with this common injury throughout the globe.

DETAILED DESCRIPTION:
Chest injuries are common in patients with polytrauma and are responsible for approximate 25% of all trauma-related mortalities. Traumatic injuries to the thorax often result in the accumulation of blood within the pleural space (i.e. a hemothorax (HTX)). The management of HTX remains a clinical dilemma when the volume of blood is small to moderate and the patient is hemodynamically stable. Prior to the ubiquitous use of chest computed tomography (CT), diagnosing quantities of blood <1000 mL was challenging (especially given inherent limitations in the standard chest radiograph (CXR)). With the widespread adoption of CT ''pan-scanning'' however, significantly more HTXs are being detected. The clinical significance and optimal treatment of these small to moderate HTXs remains unknown. Although HTXs are effectively managed with tube thoracostomy (TT) drainage of the pleural space (i.e. chest tube placement), this intervention is associated with numerous potential major complications, including iatrogenic injury, retained HTX, and empyema in up to 22% of patients. The East American Association of Trauma guidelines suggest that all HTXs should be considered for TT drainage. However, a prospective observational study suggested small to moderate HTXs could be absorbed without intervention. Classic studies from the 1960's also indicate that much larger quantities of blood can be reabsorbed without intervention as well. As a result, it is unclear if chest tubes are being over-utilized in patients who may not actually require them. Retrospective data from over 2,000 patients also suggests that many traumatic HTXs can be managed expectantly without TT drainage. Finally many small or occult HTXs (those not diagnosed by CXR, but later detected by CT scan) may also be safely observed, thus supporting the concept of expectant management (EM) for many HTXs with the goal of minimizing patient morbidity.

The Foothills Medical Centre recently reported a retrospective study including 635 patients with traumatic HTXs. Overall, 491 (66%) HTXs were drained while 258 (34%) were managed expectantly. Independent predictors of TT placement included concomitant ipsilateral flail chest or pneumothorax. It also became evident that clinical practice was not directly dependent on the specific size of the HTX. Although the adjusted odds of mortality were not significantly different between groups (OR 3.99; 95% CI 0.87-18.30; p = 0.08), TT was associated with a 47.14% (95% CI, 25.57-69.71%; p < 0.01) adjusted increase in hospital length of stay. Empyemas (n = 29) also only occurred among TT patients. The authors concluded that expectant management of traumatic HTX was associated with a shorter length of hospital stay, no empyemas, and no increase in mortality. Although EM of small HTXs appears safe and optimal, these findings must be confirmed by a larger randomized controlled trial. The purpose of this study is therefore to conduct a randomized controlled study to compare patients with traumatic HTX managed by TT or EM. Characterization of those HTXs that require pleural drainage versus those that can be managed conservatively will be optimally defined. The results from this study will inform the care of future trauma patients who present with this common injury throughout the globe.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years
2. Blunt thoracic injury
3. CT detected hemothorax

Exclusion Criteria:

1. Hemodynamic instability that is related to HTX in the judgment of the attending clinician
2. Any scenario where the clinician mandates urgent TT placement
3. Penetrating thoracic injury
4. Respiratory distress that is related to HTX in the judgment of the attending clinician
5. Chest tube already in-situ (eg. Prior to transfer of care to the FMC)
6. >24 h after admission
7. Ipsilateral flail chest fracture pattern

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The numbers of hemothoraces that require thoracic interventions. | 1 year after patient recruited in the study
  The rate of hemothoraces that require thoracic interventions in patients of both groups.

SECONDARY OUTCOMES:
The days of mechanical ventilation in intensive care unit | 30 days after patients recruited in the study
  The median length of days of mechanical ventilation needed by the patients in both groups
The days of intensive care unit stay | 30 days after patients recruited in the study
  The median length of days in ICU needed by patients in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Chad G Ball, MD, Principal Investigator — University of Calgary
Locations (2):
- Canada (2):
  - Foothills Medical Centre, Calgary, Alberta
  - Foothills Medical Centre, Faculty of Medicine, Calgary, Alberta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stafford RE, Linn J, Washington L. Incidence and management of occult hemothoraces. Am J Surg. 2006 Dec;192(6):722-6. doi: 10.1016/j.amjsurg.2006.08.033. PMID 17161082
- [Result] Ball CG, Lord J, Laupland KB, Gmora S, Mulloy RH, Ng AK, Schieman C, Kirkpatrick AW. Chest tube complications: how well are we training our residents? Can J Surg. 2007 Dec;50(6):450-8. PMID 18053373
- [Result] DuBose J, Inaba K, Okoye O, Demetriades D, Scalea T, O'Connor J, Menaker J, Morales C, Shiflett T, Brown C, Copwood B; AAST Retained Hemothorax Study Group. Development of posttraumatic empyema in patients with retained hemothorax: results of a prospective, observational AAST study. J Trauma Acute Care Surg. 2012 Sep;73(3):752-7. doi: 10.1097/TA.0b013e31825c1616. PMID 22929504
- [Result] Bradley M, Okoye O, DuBose J, Inaba K, Demetriades D, Scalea T, O'Connor J, Menaker J, Morales C, Shiflett T, Brown C. Risk factors for post-traumatic pneumonia in patients with retained haemothorax: results of a prospective, observational AAST study. Injury. 2013 Sep;44(9):1159-64. doi: 10.1016/j.injury.2013.01.032. Epub 2013 Feb 19. PMID 23433600
- [Result] DuBose J, Inaba K, Demetriades D, Scalea TM, O'Connor J, Menaker J, Morales C, Konstantinidis A, Shiflett A, Copwood B; AAST Retained Hemothorax Study Group. Management of post-traumatic retained hemothorax: a prospective, observational, multicenter AAST study. J Trauma Acute Care Surg. 2012 Jan;72(1):11-22; discussion 22-4; quiz 316. doi: 10.1097/TA.0b013e318242e368. PMID 22310111
- [Result] Mowery NT, Gunter OL, Collier BR, Diaz JJ Jr, Haut E, Hildreth A, Holevar M, Mayberry J, Streib E. Practice management guidelines for management of hemothorax and occult pneumothorax. J Trauma. 2011 Feb;70(2):510-8. doi: 10.1097/TA.0b013e31820b5c31. No abstract available. PMID 21307755
- [Result] Khandhar SJ, Johnson SB, Calhoon JH. Overview of thoracic trauma in the United States. Thorac Surg Clin. 2007 Feb;17(1):1-9. doi: 10.1016/j.thorsurg.2007.02.004. PMID 17650692
- [Result] Kulshrestha P, Munshi I, Wait R. Profile of chest trauma in a level I trauma center. J Trauma. 2004 Sep;57(3):576-81. doi: 10.1097/01.ta.0000091107.00699.c7. PMID 15454805
- [Result] Bilello JF, Davis JW, Lemaster DM. Occult traumatic hemothorax: when can sleeping dogs lie? Am J Surg. 2005 Dec;190(6):841-4. doi: 10.1016/j.amjsurg.2005.05.053. PMID 16307931
- [Result] Wells BJ, Roberts DJ, Grondin S, Navsaria PH, Kirkpatrick AW, Dunham MB, Ball CG. To drain or not to drain? Predictors of tube thoracostomy insertion and outcomes associated with drainage of traumatic hemothoraces. Injury. 2015 Sep;46(9):1743-8. doi: 10.1016/j.injury.2015.04.032. Epub 2015 May 7. PMID 25983221
- [Derived] Carver DA, Bressan AK, Schieman C, Grondin SC, Kirkpatrick AW, Lall R, McBeth PB, Dunham MB, Ball CG. Management of haemothoraces in blunt thoracic trauma: study protocol for a randomised controlled trial. BMJ Open. 2018 Mar 3;8(3):e020378. doi: 10.1136/bmjopen-2017-020378. PMID 29502092